CLINICAL TRIAL: NCT04725604
Title: Real-time Soft Tissue Assessment Using a Technologically Advanced pH
Brief Title: Real-time Soft Tissue Assessment Using a Technologically Advanced pH Monitoring System
Acronym: SoftpH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government); Softcell Medical Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3-061-18; 21-NS-0005 (Other: Research Ethics Committee reference)
Record Dates: First submitted 2020-12-16; First posted 2021-01-27 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Acute Compartment Syndrome
Keywords: Acute Compartment Syndrome; Fasciotomy

STUDY DESIGN:
Intervention Model Description: Blinded diagnostic field study
Masking Description: All participants will take part in pH probe monitoring. Results from the monitoring system will not be available until results are reviewed. No clinical decisions will be made using the new pH probes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pH Probe (Experimental): Softcell pH monitoring system: designed to measure intramuscular pH levels in patients with fracture or crush injuries sufficiently severe to be at risk of developing ACS.
  Interventions: Device: pH probe

INTERVENTIONS:
Device: pH probe — Patients who agree to take part will have a pH probe inserted into their injured limb. The pH probe will be attached to a pH monitor which will record pH data for up to a maximum of 72 hours (24 hours per probe). The surgical team will not have access to the pH data. During the time they are considered "at risk" for ACS, patients will be monitored in the routine way (using regular clinical assessment and pressure monitoring). If ACS is diagnosed in the routine way, then treatment (fasciotomy) will be offered as appropriate.

SUMMARY:
Acute Compartment Syndrome (ACS) can occur when there is a gradual reduction in the blood supply to injured limbs, most commonly after fractures or crush injuries. If ACS is not diagnosed early enough, it can result in muscle and other tissues dying off because of the lack of blood supply. Diagnosing ACS remains a challenge for doctors - currently clinical assessment and pressure probes are used to assess patients at risk of ACS. Previous research has shown that measuring pH in injured muscles is promising in diagnosing ACS and may help doctors diagnose ACS earlier than they can using current methods.

In this study, the investigators will use a pH probe to measure muscle pH, and in particular, any build-up of acid caused by reduced blood flow in the injured limb. The investigators will compare the pH probe values with the existing methods for diagnosing ACS.

Patients with a fracture or crush injury who are risk of developing ACS will be recruited into the study. Participants will have a pH probe inserted into tissue close to their injury and pH data will be logged for up to 72 hours. Diagnosis and any treatment decisions for participants in the study will be made using the existing methods and not based on information from the pH probe (the team treating the patient will not have access to the pH data). Data on diagnosis and any treatment given for ACS will be collected from participant's medical notes. The Soft pH trial team will compare how well the pH probe performs in diagnosing ACS compared to the existing methods. The investigators will follow participants up at 6 months after their initial injury to identify missed ACS cases based on clinical findings.

Diagnosing ACS earlier may reduce the likelihood of long-term symptoms and loss of function that is often seen in cases of ACS.

DETAILED DESCRIPTION:
Patients who are admitted to an orthopaedic trauma unit or intensive care unit with fractures or crush injuries and who are at risk of developing Acute Compartment Syndrome (ACS) are eligible for the study.

These patients will undergo routine monitoring for signs and symptoms of ACS. Patients who are able to make decisions about the ongoing treatment of their injured limb will be approached about the study. The patient will initially be given a short verbal statement about the study. At this point, patients may agree to take part or request additional information about the study. If patients request additional information, they can be offered a brief Patient Information Leaflet (PIL) or more detailed PIL. After reading this, they may agree to take part. Patients who agree to take part can either give verbal agreement to take part at this stage, or written informed consent.

Patients who agree to take part will have a pH probe inserted into their injured limb. The pH probe will be attached to a pH monitor which will record pH data for up to a maximum of 72 hours (24 hours per probe). The surgical team will not have access to the pH data. During the time participants are considered "at risk" for ACS, patients will be monitored in the routine way (using regular clinical assessment and pressure monitoring). If ACS is diagnosed in the routine way, then treatment (fasciotomy) will be offered as appropriate.

Once patients start to recover, written informed consent will be sought from those participants who gave verbal agreement at the outset of their participation in the study.

Until their discharge from hospital, clinical information will be collected from their medical notes or collected directly onto the study case report forms. Information from the pH monitor will be downloaded into the study website.

Participants will usually be followed up as part of routine care approximately 6 months after their initial injury. Where possible, the study follow-up will coincide with this routine follow-up. The study follow-up will include clinical examination of the limb that sustained the initial injury (including any evidence of contracture, strength of flexion/extension and any sensory abnormalities). At the 6 month follow-up participants will also be asked to complete a quality of life questionnaire.

The primary objective is to establish that the Softcell pH monitoring system measures muscle pH in an injured limb over time, monitoring changes in muscle pH that are consistent with ischaemia (drops in pH).

The properties of the pH probe as a diagnositic test will be investigated. The first analysis will be carried out after recruitment is complete, and initial data (up to 72 hours monitoring for ACS, and to potential discharge) is available. For this analysis, the presence of disease will be defined as fasciotomy within 72 hours.

A second analysis will be undertaken at the end of the study after the 6 month patient reviews have been undertaken. For this analysis, the presence of disease will be defined as fasciotomy within 72 hours OR evidence of contracture at 6 months OR significant reduction in strength OR significant sensory loss which is not improving by six months that anatomically suggest ACS.

ELIGIBILITY:
Inclusion Criteria:

* Orthopaedic Limb injuries that are at increased risk of developing ACS. In particular the following injuries will have been sustained to permit inclusion:

  1. Tibial diaphyseal fractures
  2. High energy injuries around the knee (such as dislocations of the knee, fracture dislocations of the knee or complex fractures involving the proximal tibia e.g. Shatzker IV - VI types).
  3. Forearm diaphyseal fractures
  4. High energy injuries around the elbow resulting in complex fracture dislocations.
  5. Significant crush injuries to the lower or upper limbs, including thigh, lower leg, upper arm and forearm, where compartment syndrome is suspected, in the presence or absence of a fracture.
* Male and female participants will be a minimum of sixteen years of age and under 60 years of age.
* Participants should be able to understand spoken and written English.
* Able and willing to give verbal agreement or informed consent to participate.

Exclusion Criteria:

* Patients who have evidence of previous ACS in the affected limb are not eligible.
* Patients who were, prior to injury, receiving anticoagulant therapy (with the exception of aspirin or other anti-platelet aggregation drugs) for pre-existing conditions should also be excluded from the study.
* Patients who have other illnesses/disease processes for whom the study could be detrimental will be excluded from the study (for example those with blood clotting disorders, current leukaemia, currently chemotherapy treatment, visible signs of peripheral vascular disease).
* Eligible patients will have recently sustained a serious injury - in these circumstances, pregnancy testing is challenging and not routinely done in clinical practice. We will exclude patients who declare that they are pregnant.

Ages: 16 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-07-28 (Estimated); Study Completion 2025-07-28 (Estimated)

PRIMARY OUTCOMES:
Intra-muscular pH | up to 72 hours
  ph measured by Softcell device

SECONDARY OUTCOMES:
Intra-compartmental pressure | up to 72 hours
  pressure as measured by standard clinical equipment
No of people with Acute Compartment Syndrome | Up to 72 hours
  Standard clinical assessment for Acute Compartment Syndrome up to 72 hours
No of people with Acute Compartment Syndrome | At 6 months
  Standard clinical assessment for Acute Compartment Syndrome at 6 months
Generic Quality of Life | 6 months
  EQ-5D-5L Scored -10 -100. (-10 being the worst health you can imagine and 100 being the best health you can imagine
Disease specific Quality of Life - Upper limb | 6 months
  Disabilities of the Arm, Shoulder and Hand - Scored from 0 - 100 (0 = no disability , 100 = severely disabled)
Disease specific Quality of Life - Lower limb | 6 months
  Short Musculoskeletal Function Assessment - Scored from 0 - 100 (o = no disability, 100 = severely disabled).
Number of participants with adverse events | Up to 144 hours
  Standard clinical assessment for adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Iain Stevenson, Principal Investigator — NHS Grampian
Locations (7):
- United Kingdom (7):
  - NHS Grampian, Aberdeen, Aberdeen City
  - University Hospital Birmingham, Birmingham
  - NHS Tayside, Dundee
  - NHS Lothian, Edinburgh
  - NHS Greater Glasgow and Clyde - Glasgow Royal Infirmary, Glasgow
  - NHS Greater Galsgow and Clyde - Queen Elizabeth University Hospital, Glasgow
  - NHS Greater Glasgow and Clyde - Royal Alexandra Hospital, Glasgow

IPD SHARING:
Plan to Share IPD: No